CLINICAL TRIAL: NCT01171118
Title: Phamacological Reversal of Airway Instability During Sedation
Acronym: PHYSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Suzanne Karan, Principal investigator, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17789
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Upper Airway Obstruction
Keywords: Breathing; Sedation
MeSH Terms: conditions — Airway Obstruction; Respiratory Aspiration | interventions — Physostigmine; physostigmine salicylate; Oxygen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sedation & Physostigmine & Room Air (Experimental): We are attempting to demonstrate a decrease in the frequency and severity of sedation-induced respiratory arrhythmias (central and obstructive apneas) with pharmacological pre-treatment in this pilot project and then eventually to understand the mechanisms behind this decrease. The efficacy and mechanisms of these treatments, while evaluated during sleep in OSA patients, have not been systematically studied during sedation in either normal subjects or OSA patients. The agent to be assessed in this study is physostigmine versus placebo.We are interested in the effect of breathing oxygen vs. room air on the regulation of respiratory control during moderate sedation.
  Interventions: Drug: Physostigmine
- Sedation & Placebo & Room Air (Placebo Comparator): We are attempting to demonstrate a decrease in the frequency and severity of sedation-induced respiratory arrhythmias (central and obstructive apneas) with pharmacological pre-treatment in this pilot project and then eventually to understand the mechanisms behind this decrease. The efficacy and mechanisms of these treatments, while evaluated during sleep in OSA patients, have not been systematically studied during sedation in either normal subjects or OSA patients. The agent to be assessed in this study is physostigmine versus placebo.We are interested in the effect of breathing oxygen vs. room air on the regulation of respiratory control during moderate sedation.
  Interventions: Drug: Placebo
- Sedation & Physostigmine & Oxygen (Experimental): We are attempting to demonstrate a decrease in the frequency and severity of sedation-induced respiratory arrhythmias (central and obstructive apneas) with pharmacological pre-treatment in this pilot project and then eventually to understand the mechanisms behind this decrease. The efficacy and mechanisms of these treatments, while evaluated during sleep in OSA patients, have not been systematically studied during sedation in either normal subjects or OSA patients. The agent to be assessed in this study is physostigmine versus placebo.We are interested in the effect of breathing oxygen vs. room air on the regulation of respiratory control during moderate sedation.
  Interventions: Drug: Physostigmine; Drug: Oxygen
- Sedation & Placebo & Oxygen (Placebo Comparator): We are attempting to demonstrate a decrease in the frequency and severity of sedation-induced respiratory arrhythmias (central and obstructive apneas) with pharmacological pre-treatment in this pilot project and then eventually to understand the mechanisms behind this decrease. The efficacy and mechanisms of these treatments, while evaluated during sleep in OSA patients, have not been systematically studied during sedation in either normal subjects or OSA patients. The agent to be assessed in this study is physostigmine versus placebo.We are interested in the effect of breathing oxygen vs. room air on the regulation of respiratory control during moderate sedation.
  Interventions: Drug: Oxygen; Drug: Placebo

INTERVENTIONS:
Drug: Physostigmine — Physostigmine is a centrally acting acetylcholinesterase inhibitor that has been proposed as a treatment for sleep disordered breathing. It is currently FDA approved and used commonly by Anesthesiologists in the post anesthetic setting to reverse confusion caused by central anticholinergic medication effects.
  Other Names: Antilirium
  Arms: Sedation & Physostigmine & Oxygen; Sedation & Physostigmine & Room Air
Drug: Oxygen — The administration of nasal cannula-administered oxygen at a flow rate of 2 liters/minute is commonly performed during clinical sedation practice. Thus, this experiment employed its use to compare respiratory effects of oxygen versus room air.
  Arms: Sedation & Physostigmine & Oxygen; Sedation & Placebo & Oxygen
Drug: Placebo — The administration of placebo versus physostigmine was untertaken in the same sedation conditions on the alternate day in each subject (and with both room air and oxygen)
  Other Names: Normal Saline
  Arms: Sedation & Placebo & Oxygen; Sedation & Placebo & Room Air

SUMMARY:
The investigators are attempting to demonstrate a decrease in the frequency and severity of sedation-induced respiratory arrhythmias(central and obstructive apneas) with pharmacological pre-treatment in this pilot project and then eventually to understand the mechanisms behind this decrease. The efficacy and mechanisms of these treatments, while evaluated during sleep in Obstructed Sleep Apnea (OSA) patients, have not been systematically studied during sedation in either normal subjects or OSA patients. The agent to be assessed in this study in physostigmine versus placebo.

DETAILED DESCRIPTION:
One of the most serious side effects of drugs administered for sedation is untoward respiratory events. The relative prevalence of such events is thought to be high, occurring in up to 41% of patients in some cohorts. Many specific drugs and combinations have been recommended for moderate sedation, particularly when provided by a non-anesthesiologist. The use of an opioid and a benzodiazepine is the most frequent combination, partly because the availability of antagonists for both drugs may make a "rescue" easier. However, this combination results in frequent respiratory arrhythmias (combinations of obstructions, pauses and changes in respiratory patterns).There has not been a comprehensive study of the mechanisms underlying the disruptions of respiratory rhythm caused by agents commonly used for moderate sedation. This specific research, and the line of research it opens, has the potential to make the administration of anxiolytics and analgesics safer for patients at high risk for respiratory events.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45
* BMI below 25
* Healthy males

Exclusion Criteria:

* Psychiatric illness
* Substance abuse
* Airway disorders
* Bleeding abnormatlities
* Claustrophobia
* Sleep apnea.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne B Karan, Medical, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment August 2009 to December 2010. Subjects were recruited from advertisements.
Pre-assignment Details: Subjects excluded from trial before assignment to group because BMI to high, medication exclusions, lost of follow up, scheduling conflict.
Groups:
- Physostigmine vs. Placebo in Room Air vs. O2 During Sedation: Each subject received the sedation protocol as described below:
  Midazolam : The sedation will be initated with a midazolam infusion with an effect-site target of 100 mg/ml intraventously Remifentanil : 0.3 mg/ml intravenously continuously Then, subjects were randomized to the specific order of each four arms. Physostigmine (PS) vs. Placebo were randomized by DAYS. Then, on each day, subjects were randomized to receive oxygen or room air first or second. But each subject went through BOTH days and both oxygen and room air on each day.
  There were eight total possible sequences.
Period: Overall Study
Arm/Group | Physostigmine vs. Placebo in Room Air vs. O2 During Sedation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 10 subjects were studied in a crossover format but each subject completed all arms of the study.
Groups:
- Physostigmine/Placebo: Physostigmine (PS), a centrally-acting acetylcholinesterase inhibitor, is most commonly used by anesthesiologists in the post-anesthetic setting to reverse confusion caused by central anticholinergic medication effects. It has also been proposed as a treatment for sleep disordered breathing.We investigated whether PS was effective in decreasing the frequency of ventilatory arrhythmias (VA) produced during moderate sedation with midazolam and remifentanil in both room air (RA) and 2 l/m nasal O2. Midazolam : The sedation will be initated with a midazolam infusion with an effect-site target of 100 mg/ml intraventously Remifentanil : 0.3 mg/ml intravenously continuouslyCapsaicin : 0.075% topical cream applicationPlacebo:We are attempting to demonstrate a decrease in the frequency and severity of sedation-induced respiratory arrhythmias (central and obstructive apneas) with pharmacological pre-treatment in this pilot project and then eventually to understand the mechanisms behind this.
Arm/Group | Physostigmine/Placebo
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: AHI - Apnea Hypopnea Index
Description: This is a standard metric used to describe severity of disordered breathing during sleep.Normal healthy subjects would have an AHI value of zero during sleep. Mild disordered breathing would correspond to a value of 5 to 10 events per hours; moderate 10-25; severe would be over 25
Time Frame: 2- 2 1/2 hours during study visit
Population: This is a standard size for this type of sleep study and was performed per protocol.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Physostigmine/Oxygen; Placebo/Oxygen: Physostigmine (PS), a centrally-acting acetylcholinesterase inhibitor, is most commonly used by anesthesiologists in the post-anesthetic setting to reverse confusion caused by central anticholinergic medication effects. It has also been proposed as a treatment for sleep disordered breathing.We investigated whether PS was effective in decreasing the frequency of ventilatory arrhythmias (VA) produced during moderate sedation with midazolam and remifentanil in both room air (RA) and 2 l/m nasal O2. Midazolam : The sedation will be initated with a midazolam infusion with an effect-site target of 100 mg/ml intraventously Remifentanil : 0.3 mg/ml intravenously continuously Capsaicin : 0.075% topical cream application Subjects were breathing oxygen via nasal cannula at 2 liters/minute
- Physostigmine/Room Air; Placebo/Room Air: Each subject received the sedation protocol as described below:
  Midazolam : The sedation will be initated with a midazolam infusion with an effect-site target of 100 mg/ml intraventously Remifentanil : 0.3 mg/ml intravenously continuously Then, subjects were randomized to the specific order of each four arms. Subjects breathed room air and received placebo instead of physostigimine in this arm.
Arm/Group | Physostigmine/Oxygen | Placebo/Oxygen | Physostigmine/Room Air | Placebo/Room Air
Number analyzed (Participants) | 10 | 10 | 10 | 10
events per hour | 14.5 (21.7) | 27.9 (49.3) | 11.3 (19.4) | 12.1 (21.1)

ADVERSE EVENTS:
Groups:
- Physostigmine: Physostigmine (PS), a centrally-acting acetylcholinesterase inhibitor, is most commonly used by anesthesiologists in the post-anesthetic setting to reverse confusion caused by central anticholinergic medication effects. It has also been proposed as a treatment for sleep disordered breathing.We investigated whether PS was effective in decreasing the frequency of ventilatory arrhythmias (VA) produced during moderate sedation with midazolam and remifentanil in both room air (RA) and 2 l/m nasal O2. Midazolam : The sedation will be initated with a midazolam infusion with an effect-site target of 100 mg/ml intraventously Remifentanil : 0.3 mg/ml intravenously continuously Capsaicin : 0.075% topical cream application
- Placebo: We are attempting to demonstrate a decrease in the frequency and severity of sedation-induced respiratory arrhythmias (central and obstructive apneas) with pharmacological pre-treatment in this pilot project and then eventually to understand the mechanisms behind this decrease. The efficacy and mechanisms of these treatments, while evaluated during sleep in OSA patients, have not been systematically studied during sedation in either normal subjects or OSA patients. The agent to be assessed in this study is physostigmine versus placebo.
- Oxygen: Subjects were assessed for two separate one hour periods of time -- one hour while breathing oxygen via a nasal cannula at 2 liters/minute
- Room Air: Subjects were assessed for two separate one hour periods of time -- one hour while breathing room air
Arm/Group | Physostigmine | Placebo | Oxygen | Room Air
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Study done on healthy non OSA male patients. Has to be confirmed with patients suffering from moderate to severe OSA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes